CLINICAL TRIAL: NCT06132737
Title: An Open-label Dose Escalation Study to Evaluate Safety, Tolerability, Biodistribution and Efficacy of [90Y]Y-PentixaTher for the Therapy of Recurrent or Refractory Primary or Isolated Secondary Central Nervous System Lymphoma.
Brief Title: [90Y]Y-PTT Endoradiotherapy in CNS Lymphoma Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pentixapharm AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PTT101
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: CNS Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [90Y]Y-PTT (Experimental): The study will be performed in three cohorts with different dose levels. Eligible patients will receive one cycle of 90Y-PTT, which will be administered intravenously.
  Interventions: Drug: [90Y]Y-PentixaTher

INTERVENTIONS:
Drug: [90Y]Y-PentixaTher — [90Y]Y-PTT i.v. injection
  Other Names: [90Y]Y-PTT

SUMMARY:
This will be an open-label, single-arm, national phase 1/2 therapeutic study to evaluate the safety, tolerability, and preliminary efficacy of [90Y]Y-PentixaTher ([90Y]Y-PTT) for the treatment of recurrent or refractory primary or isolated secondary central nervous system (CNS) lymphoma.

The study will be performed in three cohorts with different dose levels according to the best-of-5 dose escalation design. A safety review committee (SRC) will evaluate dose-limiting toxicities and decide about escalation and de-escalation.

Eligible patients will receive one cycle of [90Y]Y-PTT, which will be administered intravenously. There will be no comparator in this study.

Safety, biodistribution, dosimetry and efficacy will be evaluated during the core study phase (Visit 1 until Visit 5). Thereafter three follow-up (FU) visits will take place, at three-months intervals to evaluate the extent of disease.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all of the following criteria apply and are maintained at Day -2 to Day 0 (before IMP infusion):

1. Signed informed consent, by the patient or an authorized legal guardian in case the patient is temporarily not competent due to his or her disease, obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Patients of either gender aged > 18 years.
3. Body weight < 180 kg.
4. At least one measurable lymphoma manifestation in the CNS, either contrast-enhanced lesion in the brain parenchyma or measurable meningeal lesion.
5. Histologically, cytologically or radiologically confirmed relapsed/refractory primary central nervous system lymphoma (PCNSL) or relapsed/refractory secondary central nervous system lymphoma (SCNSL). Initial histologic confirmation at first diagnosis is mandatory. No peripheral lymphoma evidence is allowed.
6. Recurrent or refractory CNSL

   1. For recurrent disease, comprising new lesions or recurrent CNSL after a complete response (CR) at that site, there are no maximum number of recurrences.
   2. Refractory CNSL comprises patients with non-responding CNSL (no objective response rate (ORR), no progressive disease (PD)) to frontline therapy, or progressive disease after an initial, partial response (PR).
7. Stored stem cells with at least ≥ 2 x 106 CD34+ cells/kg of body weight.
8. If sexually active female patient of childbearing potential: patient agrees to take adequate contraceptive measures during study participation and agrees to continue use of this method for the duration of the study and for six months after the last dose.
9. Female patient without childbearing potential: documented history (e.g., tubal ligation or hysterectomy) or is post-menopausal.
10. For male patient whose partner is of child-bearing potential: patient is willing to ensure that he and his partner use effective contraception during the study and for six months after 90Y-PTT treatment.
11. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
12. Confirmed presence of CXCR4 on technically evaluable tumor lesions documented by a visually CXCR4-positive [68Ga]Ga-PentixaFor positron emission tomography (PET) scan within two months prior to enrolment in the study or during Screening.
13. Blood test results as follows:

    1. Absolute neutrophil count: > 1.0 x 109/L
    2. Hemoglobin: ≥ 8 g/dL
    3. Platelets: ≥ 75 x 109/L
    4. Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP): ≤ 3 x ULN (upper limit of normal)
    5. Serum creatinine: ≤ 2 x ULN and Cockcroft Gault calculated glomerular filtration rate (GFR) ≥ 50 mL/min
    6. Bilirubin: ≤ 3 x ULN

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria apply during screening or Day -2 to Day 0 (before IMP infusion):

1. Known or suspected hypersensitivity to study product(s) or related products.
2. Contraindication for contrast-enhanced magnetic resonance imaging (MRI) as set out in the relevant institutional guidelines (e.g., pacemaker, defibrillator, aneurysm clip, metal in the body, renal insufficiency, severe claustrophobia etc.) or contraindication for the use of gadolinium contrast for MRI.
3. Previous participation in this study. Participation is defined as signed informed consent.
4. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice). A pregnancy test will be performed at the start of the study for all female patients of childbearing potential (i.e., not surgically sterile or two years postmenopausal).
5. Male of reproductive age who or whose partner(s) is not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice).
6. Participation in any clinical study of an approved or non-approved investigational medicinal product (IMP) within the last 30 days (or ≤ 5 terminal elimination half-lives of previous IMP, whichever is longer) before screening.
7. Any disorder (e.g., active infection, unstable angina pectoris, cardiac arrhythmia (excluding atrial fibrillation and atrial flutter, uncontrolled congestive heart failure), poorly controlled hypertension, poorly controlled diabetes mellitus [HbA1c ≥ 9%], etc.) or laboratory findings, except for conditions associated with CNS lymphoma, which in the investigator's opinion might jeopardize patient's safety or compliance with the protocol.
8. Presence of active infection, or history of serious infection six weeks prior to IMP administration. Patients with uncontrolled human immunodeficiency virus (HIV) infection as well as acute or chronic active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection are excluded (Note: Patients on antiretroviral therapy (ART) with controlled HIV infection (defined as sufficient ART compliance, non-measurable HIV and CD4+ T helper cells > 200/Micro Liter) may be enrolled, if considered eligible for study treatment by the investigator.).
9. SCNSL with systemic involvement.
10. Chronic use (> 21 days) of immunosuppressive drugs, e.g., steroids for systemic autoimmune disease, due to previous organ transplantation, or other clinically evident form of immunodeficiency. Patients receiving only acute treatment (less than 21 days) with corticosteroids can be included.
11. Any mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study, and/or evidence of an uncooperative attitude without designated legal representative.
12. Brain radiation therapy ≤ 180 days before IMP infusion.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2027-09-23 (Estimated); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and relationship of (S)AEs (graded in severity according to NCI CTCAE version 5.0) | From screening until including the last follow-up visit. SAEs occuring after the end of the study should only be reported to Pentixapharm if the Investigator considers there is a causal relationship with the study drug.
  Incidence, severity and relationship of (/serious) adverse events (S)AEs will be analyzed by descriptive statistical methods. The analyses will be based on the safety analysis set (SAF).
  AEs as well as SAEs will be tabulated. Verbatim terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), and tabulations will occur by System Organ Class and Preferred Term. Severity will be graded and tabulated according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Treatment-emergent AEs will be the focus of the analyses. AEs and SAEs assessed as causality related to IMP by the investigator, and AEs leading to death will be tabulated separately.

SECONDARY OUTCOMES:
Maximal uptake (%) for tumor lesion | 1 ± 0.5 hours post infusion (p.i.).; 5 ± 1 hours p.i.; 22 ± 4 hours p.i.; 30 ± 4 hours p.i.
  The lesion activity values will be determined manually. Two volume of interests (VOIs) are drawn around a slightly enlarged organ/lesion contour, based on the computed tomography (CT) and a sphere centered around the maximal activity.
Maximal uptake (%) in discernible organs | 1 ± 0.5 hours post infusion (p.i.); 5 ± 1 hours p.i.; 22 ± 4 hours p.i.; 30 ± 4 hours p.i.
  The organ activity values will be determined manually. Two volume of interests (VOIs) are drawn around a slightly enlarged organ/lesion contour, based on the CT and a sphere centered around the maximal activity.
TAC in discernible thoracic and abdominal organs, target lesion and blood | Discernible thoracic /abdominal organs /target lesion: 1 ± 0.5 hours post infusion (p.i.).; 5 ± 1 hours p.i.; 22 ± 4 hours p.i.; 30 ± 4 hours p.i. For Blood: 5 ± 2 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 5 ± 1 hours, 22 ± 4 hours, 48 ± 6 hours p.i.
  The organ/lesion activity values will be determined manually. Two volume of interests (VOIs) are drawn around a slightly enlarged organ/lesion contour, based on the CT and a sphere centered around the maximal activity.
  For both evaluations the total activity will be noted and scaled to the injected activity.
  The Time activity curves (TAC) will be calculated. The blood samples will be measured in a calibrated well counter. Applying the calibration factor, the counts will be converted to activity of the blood samples.
AUC of 90Y-PTT in discernible thoracic and abdominal organs, target lesion and blood | Discernible thoracic /abdominal organs /target lesion: 1 ± 0.5 hours post infusion (p.i.).; 5 ± 1 hours p.i.; 22 ± 4 hours p.i.; 30 ± 4 hours p.i. For blood: 5 ± 2 minutes, 30 ± 5 minutes, 1 hour ± 10 minutes, 5 ± 1 hours, 22 ± 4 hours, 48 ± 6 hours p.i.
  The organ/lesion activity values will be determined manually. Two volume of interests (VOIs) are drawn around a slightly enlarged organ/lesion contour, based on the CT and a sphere centered around the maximal activity.
  For both evaluations the total activity will be noted and scaled to the injected activity.
  The time activity curves (TAC) will be calculated. The blood samples will be measured in a calibrated well counter. Applying the calibration factor, the counts will be converted to activity of the blood samples.
  The area under the curve (AUC) will be calculated.
AUC of 90Y-PTT in urine | 0 - 5 hours (before 2nd PET scan); 5 - 22 hours (before 3rd PET scan); 22 - 48 hours
  The activity concentrations of the collected urine will be measured in a well counter.
  The area under the curve (AUC) will be calculated.
Organ receiving the highest absorbed dose | 1 ± 0.5 hours post infusion (p.i).; 5 ± 1 hours p.i.; 22 ± 4 hours p.i.; 30 ± 4 hours p.i.
  The organ/lesion activity values will be determined manually. Two volume of interests (VOIs) are drawn around a slightly enlarged organ/lesion contour, based on the computed tomography (CT) and a sphere centered around the maximal activity.
Cumulative absorbed organ/lesion doses (Gy) | 1 ± 0.5 hours post infusion (p.i).; 5 ± 1 hours p.i.; 22 ± 4 hours p.i.; 30 ± 4 hours p.i.
  The organ/lesion activity values will be determined manually. Two volume of interests (VOIs) are drawn around a slightly enlarged organ/lesion contour, based on the CT and a sphere centered around the maximal activity.
ORR at one month and three months | Month 1 (Visit 4) and Month 3 (Visit 5)
  Proportion of patients who have partial response or complete response after treatment during study duration according to (International Primary Central Nervous System Lymphoma Collaborative Group) IPCG response criteria. This is also called the objective response rate (ORR).
PFS at one month and three months | Month 1 (Visit 4) and Month 3 (Visit 5) post infusion
  Proportion of patients whose status results in death or progressive disease or disease relapse after achieving complete response according to IPCG response criteria. This is also called progression-free survival (PFS).
Rate of CR and PR at one month and three months | Month 1 (Visit 4) and Month 3 (Visit 5) post infusion
  Proportion of patients with complete response (CR) and partial response (PR) according to IPCG response criteria.
PFS at 12 month (including a nine-month FU according to the local investigator's discretion) | 6 months post infusion (p.i.); 9 months p.i.; 12 months p.i.;
  Progression free survival (PFS) of patients according to IPCG response criteria.
OS at 12 month (including a nine-month FU according to the local investigator's discretion) | 6 months post infusion (p.i.); 9 months p.i.; 12 months p.i.;
  Overall survival (OS) at 6 months, 9 months and 12 months after infusion is assessed.

OTHER OUTCOMES:
Incidence and severity of DLT | Up to 28 days post infusion
  DLT (Dose limiting toxicity) is defined as a toxicity with a severity that prevents further increase in dose level.
  The incidence and the severity will be assessed.
Changes from baseline in vital signs | Baseline: -28 to -8 days before infusion; End of infusion; 5 ± 2 / 30 ± 5 minutes post infusion (p.i) ; 1 hour ± 10 minutes p.i.; 5 ± 1 / 22 ± 4 hours p.i. ; 22 to 48 hours p.i.; 2 / 14 days p.i.; 1/ 3 / 6 / 9 / 12 months p.i.
  Changes from the values of vital signs at screening visit will be assessed during the trial at different time points.
Changes from baseline in laboratory parameters (hematology and biochemistry) | Hematology/Biochemistry: -28 to -8 days before infusion; Before infusion; 5 ± 1 hours post infusion (p.i.).; 2 days p.i.; 14 ± 2 days p.i; 1 / 3 months ± 5 days p.i.; 6 / 9 / 12 months ± 14 days p.i.;
  Changes from the values of laboratory parameters will be assessed during the trial at different time points.
Changes from baseline in laboratory parameters (urinalysis) | Urinalysis: -28 to -8 days before infusion; 0 to 5 hours post infusion (p.i.) (before 2nd scan); 5 to 22 hours p.i.(before 3rd scan); 22 to 48 hours p.i.(before 4th scan); 2 days p.i.; 14 ± 2 days p.i; 1 / 3 months ± 5 days p.i.;
  Changes from the values of laboratory parameters will be assessed during the trial at different time points.
Abnormal findings in physical examination | -28 to -8 days before infusion; Before infusion; 2 days post infusion (p.i.); 14 ± 2 days p.i; 1 / 3 months ± 5 days p.i.; 6 / 9 / 12 months ± 14 days p.i.;
  Changes from values of the physical examination will be assessed during the trial at different time points.
Findings12-lead ECG | -28 to -8 days before infusion; Before infusion; 5 ± 1 hours post infusion (p.i.); 2 days p.i.; 14 ± 2 days p.i; 1 / 3 months ± 5 days p.i.
  Changes from values of the 12-lead electrocardiogram (ECG) will be assessed during the trial at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Bastian von Tresckow, Prof. Dr. med., Principal Investigator — University Hospital, Essen
Locations (2):
- Germany (2):
  - University Hospital Rechts der Isar, Munich, Bavaria
  - University Hospital Essen, Essen